CLINICAL TRIAL: NCT00512005
Title: Valvular and Ventricular Improvement Via iCoapsys Delivery (VIVID) Feasibility Study
Brief Title: VIVID - Valvular and Ventricular Improvement Via iCoapsys Delivery - Feasibility Study
Acronym: VIVID
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Myocor (Industry)
Responsible Party: Cyril J. Schweich, MD / VP of Clinical and Regulatory Affairs, Myocor, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030301
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2008-05

CONDITIONS: Mitral Valve Regurgitation; Left Ventricular Dysfunction; Heart Failure; Mitral Insufficiency; Mitral Incompetence; Ischemic Heart Disease
Keywords: Functional Mitral Regurgitation (FMR); Ischemic Mitral Regurgitation; Less invasive repair; Percutaneous MV repair; Mitral Valve Repair; Heart Failure; Left Ventricular Dysfunction
MeSH Terms: conditions — Mitral Valve Insufficiency; Ventricular Dysfunction, Left; Heart Failure; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Percutaneous mitral valve repair — Ventricular reshaping to treat functional mitral insufficiency
  Other Names: iCoapsys System

SUMMARY:
The purpose of this prospective, non-randomized, single-arm feasibility study is to evaluate safety and feasibility of the iCoapsys System in patients with functional mitral valve insufficiency caused by annular dilation and/or papillary muscle displacement.

DETAILED DESCRIPTION:
Functional MR is a frequent outcome of ischemic heart disease or dilated cardiomyopathy. Patients with functional MR generally have normal valvular structures complicated by left ventricular dysfunction. Left ventricular dysfunction will often create geometric distortions that prevent complete leaflet coaptation, rendering the valve incompetent. Changes that will induce functional MR may include (i) dyskinetic or akinetic wall segments, (ii) dilation of the valve annulus or (iii) dilation of the left ventricle leading to tethering of the chordae tendinae.

The iCoapsys Device is intended to treat patients with functional MR. The device is not indicated for patients with diseased or damaged valvular structures caused by rheumatic fever, degenerative diseases, endocarditis, infiltrative diseases or congenital disorders.

ELIGIBILITY:
Key Inclusion Criteria:

* Grade 3 or 4 functional mitral valve regurgitation per 2D echocardiography.
* NYHA Class II and LVEF greater than or equal to 25% or NYHA Class III and LVEF greater than or equal to 30%

Key Exclusion Criteria:

* History of pericarditis.
* Creatinine > 2.2 at the time of the procedure
* INR > 1.8 at the time of the procedure
* Prior pericardial intervention (including CABG, pericardiotomy or pericardiocentesis).
* Any endovascular therapeutic interventional or surgical procedure performed within 30 days prior to the index procedure (e.g., stent placement).
* Any planned therapeutic interventional or surgical procedure planned within 30 days following the index procedure
* Open chest surgery contraindication (e.g., acute respiratory distress, endocarditis, myocarditis).
* Structural abnormality of the mitral valve
* Valve disease resulting in insufficiency or stenosis of the aortic, pulmonary or tricuspid valve requiring intervention.
* Pericardial effusion >5 mm via echocardiography.
* Posterior wall end-diastolic dimension >1.3 cm.
* Left ventricular end diastolic diameter > 7.0 cm.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Intra-procedural implant safety of iCoapsys System, Peri-procedural safety of the iCoapsys System, Intra-procedural MR reduction with the iCoapsys System | Intra-procedure and peri-procedure

SECONDARY OUTCOMES:
Minnesota Living with Heart Failure Questionnaire, 6-Minute Hallwalk, LV Chamber Volumes | 1, 3, 6, 12, 18, 24 months and annually thereafter

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Emory University Hospital, Atlanta, Georgia
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Shawnee Mission Hospital, Shawnee Mission, Kansas
  - Abbott Northwestern Hospital, Minneapolis, Minnesota